CLINICAL TRIAL: NCT03926052
Title: Cognitive-Behavioral and Pharmacologic (LDX) Treatment of Binge-Eating Disorder and Obesity
Brief Title: Cognitive-Behavioral and Pharmacologic (LDX) Treatment of Binge-Eating Disorder and Obesity: Maintenance Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000022480; 1R01DK114075-01A1 (NIH)
Record Dates: First submitted 2019-04-18; First posted 2019-04-24 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Binge-Eating Disorder; Obesity
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LDX (Active Comparator)
  Interventions: Drug: Lisdexamfetamine Dimesylate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate — Participants randomly assigned to this arm will receive 12 weeks of LDX medication.
  Arms: LDX
Drug: Placebo — Participants randomly assigned to this arm will receive 12 weeks of an inactive placebo.
  Arms: Placebo

SUMMARY:
This study will test the effectiveness of lisdexamfetamine (LDX) medication as a maintenance therapy for the treatment of binge-eating disorder (BED) in patients with obesity. This is a controlled test of whether, amongst responders to acute treatments, LDX medication results in superior maintenance and longer-term outcomes compared with placebo.

DETAILED DESCRIPTION:
Obesity is a heterogeneous problem and research has highlighted the particular significance of a subgroup with binge-eating disorder (BED), the most prevalent formal eating disorder. Improved treatments for patients with obesity and BED are needed that can produce sustained clinical outcomes and promote weight loss. This study (maintenance stage) RCT will provide findings from a controlled test, amongst responders to acute treatments, whether LDX medication results in superior maintenance and longer-term outcomes than placebo. This is one of the few RCTs for BED of medication with follow-up after medication discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years old
* Meets DSM-5 criteria for binge-eating disorder
* BMI 27-30 with a controlled obesity-related co-morbidity; or BMI ≥ 30 and <50
* Medically cleared as determined by EKG and medical record review
* Available for the duration of the treatment and follow-up (18 months)
* Read, comprehend, and write English at a sufficient level to complete study-related materials
* Able to travel to study location (New Haven, CT) for weekly visits

Exclusion Criteria:

* Previous history of problems with LDX or other stimulants
* Current psychostimulant use or use of any medication for ADHD
* Current use of study medications: LDX (Vyvanse), Bupropion (Wellbutrin, Zyban), Naltrexone, or Contrave
* History of congenital heart disease, known structural cardiac abnormalities, cardiomyopathy, serious heart arrhythmia, coronary artery disease, cerebrovascular pathology including stroke, exertional chest pain, uncontrolled high blood pressure, and other serious heart problems.
* History of severe renal, hepatic, neurological, or chronic pulmonary disease or other serious, unstable medical disorder.
* Current uncontrolled hypertension
* Current uncontrolled type I or II diabetes mellitus
* Current uncontrolled thyroid illness
* Gallbladder disease
* Co-occurring severe mental illness requiring hospitalization or intensive treatment
* Endorses current active suicidal or homicidal ideation with intent or plan
* History or current alcohol or substance use disorder (smoking is not exclusionary)
* Predisposition to seizures
* History of anorexia nervosa or bulimia nervosa, or currently regularly self-inducing vomiting
* Currently taking MAOI, SSRI or strong inhibitors of CYP2D6
* History of allergy or sensitivity to the study medication or stimulant medications
* Current use of medications contraindicated with the study medications
* Currently breast feeding or pregnant, or not willing to use reliable form of contraception
* Currently taking opioid pain medications or drugs
* Currently using effective treatment (evidence-based therapeutic or psychopharmacologic) for eating and/or weight loss
* Currently participating in another clinical study in which the participant is or will be exposed to an investigational or a non-investigational drug or device
* Medical status judged by study physician as contraindication

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Grilo, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Department of Psychiatry, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LDX (Lisdexamfetamine Dimesylate): Lisdexamfetamine Dimesylate: Participants randomly assigned to this arm will receive 12 weeks of LDX medication.
Period: Overall Study
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Started | 32 | 29
Completed | 30 | 28
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.97 (11.38) | 45.83 (10.24) | 44.33 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 25 | 21 | 46
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 32 | 29 | 61

OUTCOME MEASURES:

1. Primary Outcome: Binge-Eating Relapse
Description: Relapse will be scored as a yes/no (categorical variable); this categorical variable will be based on frequency of binge-eating episodes assessed using the Eating Disorder Examination interview; Relapse category will be defined as ≥4 binge-eating episodes per month.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 30 | 28
Participants | 3 | 5

2. Primary Outcome: Binge-Eating Relapse
Description: as for outcome 1
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 20 | 23
Participants | 6 | 6

3. Primary Outcome: Binge-Eating Relapse
Description: as for outcome 1
Time Frame: 12 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 18 | 23
Participants | 3 | 2

4. Secondary Outcome: Change in Binge-Eating Frequency
Description: Binge-eating frequency is a continuous variable of binge-eating episodes assessed using the Eating Disorder Examination interview; Binge-eating frequency will be based on the past 28 days and defined as binge-eating episodes per month.
Time Frame: From baseline interview at study enrollment to 3 months after the 12-week treatment
Measure: Mean (Standard Deviation); unit: episodes per the past 28 days
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 30 | 28
episodes per the past 28 days | 1.33 (5.82) | 1.61 (4.37)

5. Secondary Outcome: Change in Binge-Eating Frequency
Description: as for outcome 4
Time Frame: From post-treatment to the 6-month follow-up
Measure: Mean (Standard Deviation); unit: episodes per the past 28 days
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 20 | 24
episodes per the past 28 days | 2.45 (5.39) | 1.00 (6.86)

6. Secondary Outcome: Change in Binge-Eating Frequency
Description: as for outcome 4
Time Frame: From post-treatment to the 12-month follow-up
Measure: Mean (Standard Deviation); unit: episodes per the past 28 days
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 18 | 23
episodes per the past 28 days | 1.28 (4.14) | -.09 (2.29)

7. Secondary Outcome: Change in Eating-Disorder Psychopathology (Continuous)
Description: Eating-disorder psychopathology is a continuous variable as assessed by the global score of the Eating Disorder Examination/Eating Disorder Examination-Questionnaire. Scores range from 0-6 (0=no eating-disorder psychopathology; 6=severe eating-disorder psychopathology).
Time Frame: From baseline interview at study enrollment to 3 months after the 12-week treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 28 | 27
score on a scale | -0.05 (0.77) | 0.50 (0.64)

8. Secondary Outcome: Change in Eating-Disorder Psychopathology (Continuous)
Description: as for outcome 7
Time Frame: From post-treatment to the 6-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 19 | 22
score on a scale | 0.23 (0.95) | 0.17 (0.60)

9. Secondary Outcome: Change in Eating-Disorder Psychopathology (Continuous)
Description: as for outcome 7
Time Frame: From post-treatment to the 12-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 17 | 23
score on a scale | 0.09 (0.83) | -0.07 (0.59)

10. Secondary Outcome: Change in Depressive Symptoms
Description: Depressive symptoms is a continuous variable of depressive symptomatology as assessed by the self-report measure, the Beck Depression Inventory - Second Edition. Scores range from 0-63 (0=no depressive symptoms, 63=greater depressive symptoms).
Time Frame: From baseline interview at study enrollment to 3 months after the 12-week treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 25 | 28
score on a scale | 2.16 (5.27) | 0.18 (7.07)

11. Secondary Outcome: Change in Depressive Symptoms
Description: as for outcome 10
Time Frame: From post-treatment to the 6-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 17 | 20
score on a scale | 1.12 (5.63) | 3.35 (9.14)

12. Secondary Outcome: Change in Depressive Symptoms
Description: as for outcome 10
Time Frame: From post-treatment to the 12-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 15 | 21
score on a scale | 0.07 (6.98) | 1.71 (4.95)

13. Secondary Outcome: Percent Change in Weight
Description: Negative values indicate weight loss and positive values indicate weight gain.
Time Frame: From baseline interview at study enrollment to 3 months after the 12-week treatment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 30 | 28
percent change | -2.39 (2.95) | 2.25 (2.51)

14. Secondary Outcome: Percent Change in Weight
Description: Negative values indicate weight loss and positive values indicate weight gain.
Time Frame: From post-treatment to the 6-month follow-up
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 18 | 22
percent change | 2.54 (6.32) | 0.45 (3.04)

15. Secondary Outcome: Percent Change in Weight
Description: Negative values indicate weight loss and positive values indicate weight gain.
Time Frame: From post-treatment to the 12-month follow-up
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
Number analyzed (Participants) | 17 | 23
percent change | 4.04 (6.58) | 2.67 (5.73)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | LDX (Lisdexamfetamine Dimesylate) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/29
Other Adverse Events (participants affected / at risk) | 13/32 | 6/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDX (Lisdexamfetamine Dimesylate) (N=32) | Placebo (N=29)
Decreased appetite (Gastrointestinal disorders) | 10 | 4
Dry mouth (General disorders) | 6 | 1
Insomnia (General disorders) | 6 | 4
Increased energy (General disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 3 | 1
Feeling jittery (General disorders) | 2 | 0
Increased heart rate (Nervous system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT03926052/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT03926052/ICF_000.pdf